CLINICAL TRIAL: NCT06475898
Title: Longitudinal Endpoint Assessment of Disease Burden in HD
Acronym: LEAD-HD
Status: Recruiting | Type: Observational
Sponsor: Huntington Study Group (Network)
Collaborators: University of Rochester Center for Health + Technology (Unknown); Modality.AI, Inc (Unknown); Neurotargeting LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: LEAD-HD
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
LEAD-HD is intended to collect and analyze self-reported health information from individuals with Huntington Disease (HD) or prodromal HD participating in a 24-month longitudinal natural history study using remote technologies.

DETAILED DESCRIPTION:
The LEAD-HD study will be offered via HSG's online observational research platform called myHDstory®. This direct to patient study will collect and analyze self-reported health information from individuals with Huntington Disease (HD) or prodromal HD in a 24-month longitudinal natural history study that participants complete at any time and with their own electronic device.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older;
* Be willing and able to provide informed consent electronically;
* Self-report, when answering as a participant, that you have been diagnosed with HD by a doctor, or have undergone genetic testing and been found to carry the gene mutation responsible for HD but have not been clinically diagnosed with HD (prodromal HD);
* Have the ability to answer online questions or direct someone else to enter answers for them;
* Have the ability to ambulate independently and take care of some of your personal needs;
* Have the ability to read and understand English;
* Be willing to create a unique identifier based on personal demographic information;
* Reside in the United States or its territories. Surveys can only be completed in the US. If you move outside of the US, you will no longer be able to participate;
* Own or have access to an electronic device and secure internet connectivity

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must self-report they have been diagnosed with HD by a doctor or have undergone genetic testing, been found to carry the expanded allele responsible for HD and have no clinical diagnosis (prodromal HD) (HD-ISS Stage 2 or 3).
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
PRO natural history | December 2026
  Obtain PRO natural history data in HD.
Demographic characteristics | December 2026
  Identify demographic characteristics that are associated with faster or slower disease progression.
Assess the ability to consent and enroll | December 2026
  Assess the ability to consent and enroll participants in long-term longitudinal studies in HD using a direct-to-patient platform.

CONTACTS AND LOCATIONS:
Overall Officials: Jamison Seabury, Principal Investigator — University of Rochester Center for Health + Technology
Locations (1):
- Huntington Study Group, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The accrued data will help create a patient-reported natural history of HD, clinically meaningful outcomes for clinical trials, a resource to enable respondents to participate in future research, and a shared longitudinal database for researchers to access and analyze de-identified data and publish findings.
Time Frame: 2026